CLINICAL TRIAL: NCT01972646
Title: Predictors of Failure of Empiric Outpatient Antibiotic Therapy in Emergency Department Patients With Uncomplicated Cellulitis.
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Shelley McLeod, Research Program Manager, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 16936e
Record Dates: First submitted 2013-10-22; First posted 2013-10-30 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Uncomplicated Outpatient Cellulitis
Keywords: Cellulitis, treatment failure, skin and soft tissue infections, risk factors.
MeSH Terms: conditions — Cellulitis; Soft Tissue Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult patients (≥ 18 years) with uncomplicated cellulitis: Adult patients (≥ 18 years) whose chief complaint was consistent with a skin or soft tissue infection (key words included cellulitis, abscess, infection, insect bite, ulcer, or rash) were screened for eligibility by ED staff or trained research assistants and invited to participate in this study once an emergency physician confirmed a cellulitis infection.

SUMMARY:
Introduction: Despite several expert panel recommendations and cellulitis treatment guidelines, there are currently no clinical decision rules to assist clinicians in deciding which emergency department (ED) patients should be treated with oral antibiotics and which patients require intravenous therapy at first presentation of uncomplicated cellulitis. The objective of this prospective study is to determine potential patient risk factors associated with adult patients (>17years) presenting to the ED with a concern about a skin or soft tissue infection who fail initial antibiotic therapy for the treatment of standard cellulitis and require a change of antibiotics or admission to hospital.

Methods: This study will be a prospective study conducted in two tertiary care EDs. Patients will be excluded if they have been treated with antibiotics for the current bout of cellulitis prior to presenting to the ED, patients admitted to hospital and those patients with abscesses only. Hired research assistants (RAs) will administer a questionnaire at the initial ED visit with telephone follow-up 2 weeks later. Treatment failure will be defined as patients requiring subsequent hospitalization, initiation of intravenous antibiotics (if oral antibiotics were prescribed initially), or a change of oral antibiotics for the original cellulitis.

Results: This study will provide a detailed profile of patient risk factors associated with treatment failure of cellulitis. The results will be analyzed and used in formulating a clinical decision rule for effective treatment of cellulitis presenting to the ED. Each of the predictor variables associated (p ≤ 0.1) with failed treatment in the univariate analysis will be considered in a multivariate logistic regression model. Additionally, treatment variability among clinicians in regard to cellulitis will be evaluated and compared to treatment failures, thus providing data on successful treatment regimens.

Conclusions: Results from this research may be used to generate a clinical prediction rule to assist clinicians in effectively treating patients presenting to emergency departments with cellulitis. Understanding which patient risk factors for treatment failure will assist clinicians in determining which patients will benefit from intravenous versus oral antibiotics.

ELIGIBILITY:
Inclusion Criteria: Adult patients (≥ 18 years) whose chief complaint was consistent with a skin or soft tissue infection (key words included cellulitis, abscess, infection, insect bite, ulcer, or rash) were screened for eligibility by ED staff or trained research assistants and invited to participate in this study once an emergency physician confirmed a cellulitis infection.

Exclusion Criteria: Patients were excluded if they were currently taking or had been recently treated with antibiotics for the cellulitis prior to presenting to the ED, if they were admitted to hospital, had an abscess only, were cognitively impaired or did not read or speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years) whose chief complaint was consistent with a skin or soft tissue infection (key words included cellulitis, abscess, infection, insect bite, ulcer, or rash) were screened for eligibility by ED staff or trained research assistants and invited to participate in this study once an emergency physician confirmed a cellulitis infection.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
risk factors independently associated with failure of empiric outpatient antibiotic therapy in ED patients with uncomplicated cellulitis. | 16 months
  The primary objective of this study was to determine risk factors independently associated with failure of empiric outpatient antibiotic therapy in ED patients with uncomplicated cellulitis.

SECONDARY OUTCOMES:
antibiotic prescribing practices for uncomplicated cellulitis at our institution. | 16 months
  Secondary objectives were to describe the antibiotic prescribing practices for uncomplicated cellulitis at our institution.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McRae, MD, FRCPC, PhD, Principal Investigator — The University of Western Ontario
Locations (1):
- The University of Western Ontario, London, Ontario, Canada